CLINICAL TRIAL: NCT02425865
Title: Intensive Treatment to Reach the Target With Golimumab in ulcErative coliTis- In-TARGET
Brief Title: Intensive Treatment to Reach the Target With Golimumab in ulcErative coliTis - In-TARGET
Acronym: In-TARGET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2015-05
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: ULCERATIVE COLITIS
Keywords: UC, IBD
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open-label, uncontrolled trial (Other): All patients will receive Standard regimen with golimumab 50 mg Q4W, or 100 mg Q4W if > 80 kg
  Interventions: Drug: GOLIMUMAB

INTERVENTIONS:
Drug: GOLIMUMAB — Increase/ or Decrease/ Interruption Dose of Golimumab depending on Continuous Clinical Response or Relapse

SUMMARY:
PHASE: IV

TYPE OF STUDY: With direct benefit

DESCRIPTIVE: multicenter, open-label, uncontrolled trial

INCLUSION CRITERIA: Adults with moderate to severe ulcerative colitis who failed corticosteroids and immunosupressive therapy, or are intolerant to immunosuppressors. All included patients will be naïve to anti-TNF therapy. Active disease at golimumab treatment initiation defined as a MAYO score ≥6 and with an endoscopic sub score ≥2.

OBJECTIVE: To determine the proportion of patients with Continuous Clinical Response (CCR) and endoscopic remission after one year of golumimab at week 54.

STUDY DESIGN:

Induction Phase :

Week 0: golimumab 200mg- Week 2: golimumab 100 mg- Week 6: golimumab 50 mg

Maintenance Phase I : Week 10-Week 54 Week 10-Week 54 • Patients with primary clinical response*: Standard regimen with golimumab 50 mg Q4W (or 100 mg Q4W if > 80 kg)

* Patients without primary clinical response at week 10 or with flare between week 10-week 54*: Optimization to 100 mg Q4W (or combination therapy with azathioprine if > 80 kg or switch from azathioprine to methotrexate if already on azathioprine at golimumab initiation or patient with known intolerance to thiopurines)
* Early escape at Week 18: Primary non-responders who are still not responding at week 18 to dose optimization at Weeks 10 and 14 will be considered treatment failures and will be followed up (call or visit) at week 54 for safety.

  * Clinical response is defined as a decrease from baseline in the Mayo score ≥30% and ≥3 points, accompanied by either a rectal bleeding sub score of 0 or 1 or a decrease from baseline in the rectal bleeding sub score ≥1

Intermittent Phase II : Week 54-Week 108

• Patients with CCR and MH at week 54 and on golimumab 50 mg every 4 weeks: Stop golimumab and continuation of thiopurines or methotrexate if on combination therapy

• Patients with CCR and MH at week 54 and on golimumab 100 mg every 4 weeks: De-escalation to 50 mg every 4 weeks and continuation of thiopurines or methotrexate if on combination therapy

• Restart/Escalate golimumab on flare (defined in section 4 of the protocol) to the phase I dose; 50 mg q4wk or 100mg q4wk (similar to the phase I regimen)

DETAILED DESCRIPTION:
NUMBER OF PATIENTS: 200 patients

INCLUSION PERIOD: 33 months

STUDY DURATION: 57 months

MAIN EVALUATION Primary endpoints

• Week 10-54: proportion of patients in CCR and with MH (endoscopic Mayo score of 0 or 1) at week 54

Data base lock, data analysis and display (publication) will happen when all included subjects have completed the 108-week visit.

SECONDARY EVALUATION

For all included patients:

* Phase II (week 54-108): proportion of patients in CCR with MH (endoscopic Mayo score of 0 or 1) at week 108, after discontinuation or dose de-escalation (from 100 to 50 mg) of golimumab treatment at year 1 in the subgroup of patients in CCR and with MH (endoscopic Mayo score of 0 or 1) at week 54
* Factors associated with treatment success (see primary endpoint)
* Efficacy of dose optimization in patients who loose response between week 10 and 54
* Clinical remission at week 54 • Clinical remission at week 108 • Partial MAYO score at week 54 and 108 • PRO2 (Partial Mayo minus PGA) at week 54 and 108 • CCR between study inclusion and week 54 and 108 • Steroid-free clinical remission at week 54 and 108 • MH (endoscopic score MAYO 0-1) at week 54 and 108 • Changes in faecal calprotectin levels from baseline to week 54 and 108 • Colectomy between W0 and W54 and 108
* UC-related hospitalizations throughout the trial • Histological remission9 at W54 and 108
* PRO: Fatigue (FACIT), disability (IBD Disability index), QoL (SHS-IBD VAS)
* PK data (golimumab trough levels and antibodies against golimumab)
* Proportion of late responders being in Clinical Response from week 18 to week 54 and with MH at week 54 following treatment intensification in Maintenance Phase

For the subgroup of patients who are primary non-responders to golimumab at week 10, we will assess the efficacy of treatment optimization, including the percentage of patients achieving continuous clinical response and endoscopic remission at one year.

ELIGIBILITY:
INCLUSION CRITERIA

* Age sup 18 years and inf 75 years
* Established diagnosis of UC for at least 3 months (pancolitis, left-sided colitis, proctosigmoiditis and or proctitis are allowed).
* Adults with moderately-to-severely active UC who had an inadequate response to or failed to tolerate steroids AND thiopurines (azathioprine or 6-mercaptopurine) or adults with moderately-to-severely active UC who had no response to an adequate steroid course and starting golimumab.
* Active disease at golimumab treatment initiation defined as a partial MAYO score sup/equal 6 with an endoscopic sub score sup/equal 2.
* Patients concurrently treated with oral corticosteroids will receive a stable dose (prednisone 20 ≤mg/day for at least 2 weeks) before baseline.
* Patient has to be treated with oral 5-ASA at time of inclusion regardless of the dose if no contra-indication. If the patient is not on oral 5-ASA during the screening period, he/she should start mesalamine at 2g per day or asacol at 1.6 g per day, in the absence of contra-indication.
* Patients are allowed stable dose of thiopurines (azathioprine or 6-mercaptopurine stable dose for at least 4 weeks).
* Naïve to anti-TNF therapy, and other biologics, including anti-integrin antibodies and for all biologics known to be effective for UC (approved or investigational).
* Naïve to JAK inhibitors (approved or investigational)
* A contraceptive method during the whole study for childbearing potential female patients.

EXCLUSION CRITERIA

* Age under 18 and over 75.
* People unable to give their consent (because of their physical or mental state).
* Absence of written consent.
* Pregnancy or breastfeeding.
* Patients with severe acute colitis or patients at imminent risk for colectomy.
* History of colectomy.
* History of colonic mucosal dysplasia or adenomatous colonic polyps that are not removed.
* Screening stool study positive for enteric pathogens or Clostridium difficile toxin.
* Oral corticosteroids at a dose > 20 mg prednisone or its equivalent per day.
* Any current or previous use of cyclosporine, tacrolimus, anti-TNF therapy, and other biologics, including anti-integrin antibodies (approved or investigational), JAK inhibitors (approved or investigational), or any current or previous use of an investigational agent within 5 half-lives of that agent before the first study agent injection.
* Contraindication to anti-TNF therapy according to drug labelling:

  * Active infection.
  * Non-treated latent tuberculosis.
  * Heart failure (NYHA: Grade III and IV).
  * Malignancy during the previous 5 years.
  * Demyelinating neurological disease.
  * Should be vaccinated with attenuated live vaccines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Continuous Clinical Response and Endoscopic Remission | Week 54
  proportion of patients in CCR and with MH (endoscopic Mayo score of 0 or 1) at week 54

SECONDARY OUTCOMES:
Continuous Clinical Response and Endoscopic Remission after discontinuation or de- escalation of golimumab | Week 108
  proportion of patients maintaining continuous clinical response and endoscopic remission at week 108, after discontinuation or de-escalation of golimumab treatment at year 1 in the subgroup of patients in continuous clinical response (CCR) and with mucosal healing (endoscopic Mayo score of 0 or 1) at week 54
Efficacy of dose optimization in patients who loose response between week 10 and 54 | Week 54
  proportion of patients maintaining continuous clinical response after dose optimization in patients who loose response between week 10 and 54
Clinical remission at week 54 | week 54
  proportion of patient with clinical remission (partial Mayo score) at week 54
Clinical remission at week 108 | week 108
  proportion of patient with clinical remission (partial mayo score) at week 108
PRO2 (Partial Mayo minus PGA) at week 54 and 108 | week 108
  Evolution of PRO2 (Partial Mayo minus PGA) at week 54 and 108 according the clinical and endoscopic remission
CCR between study inclusion and week 54 and 108 | week 108
  proportion of patient with CCR at week 54 and 108
Steroid-free clinical remission at week 54 and 108 | week 108
  proportion of patient with steroid-free clinical remission at week 54 and 108
MH (endoscopic score MAYO 0-1) at week 54 and 108 | week 108
  proportion of patient with MH (endoscopic score MAYO 0-1) at week 54 and 108
Changes in faecal calprotectin levels from baseline at week 54 and 108 | week 108
  Evolution of faecal calprotectin levels from baseline at week 54 and 108 according the clinical and endoscopic remission
Colectomy between W0 and W54 and 108 | week 108
  Proportion of patient with colectomy between W0 and W54 and W108
UC-related hospitalizations throughout the trial | week 108
  Proportion of patient with UC-related hospitalizations throughout the trial
Histological remission at W54 and 108 | week 108
  Proportion of patient with histological remission at W54 and W108
PRO: Fatigue (FACIT), disability (IBD Disability index), QoL (SHS-IBD VAS) | week 108
  Evolution of PRO: Fatigue (FACIT), disability (IBD Disability index), QoL (SHS-IBD VAS) according the clinical and endoscopic remission
PK data (golimumab trough levels and antibodies against golimumab) | week 108
  Evolution of PK (golimumab trough levels and antibodies against golimumab) according the clinical and endoscopic remission
Late responders being in Clinical Response from week 18 to week 54 and with MH at week 54 following treatment intensification in Maintenance Phase | week 108
  Proportion of late responders being in Clinical Response from week 18 to week 54 and with MH at week 54 following treatment intensification in Maintenance Phase

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Peyrin Biroulet, MD,PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Lucine Vuitton, MD, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Edouard Louis, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (23):
- Belgium (2):
  - CHU LIEGE - Sart Tilman, Liège
  - CHU Dinant Godinne UCL Namur, Namur
- France (21):
  - CHU Amiens, Amiens
  - Chu Besancon, Besançon
  - Caen Unversity Hospital, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - APHP- Hopital BEAUJON, Clichy
  - CHU de Colmar- Hopital Trousseau Medecine A, Colmar
  - CHRU Lille, Lille
  - CHU de Montpellier- Hopital saint Eloi, Montpellier
  - CHU NANTES - Hôpital Hôtel Dieu, Nantes
  - CHU de NICE- Hopital Archet 2, Nice
  - CHU de Nimes- Hopital Carémeau, Nîmes
  - APHP- Hopital BICHAT, Paris
  - CHU Bordeaux- Hopital Haut Levèque, Pessac
  - CHU LYON- Hopital Lyon Sud, Pierre-Bénite
  - Chu Reims, Reims
  - CHU RENNES - Hopital Pontchaillou, Rennes
  - CHU de Saint Etienne- Hopital Nord, Saint-Priest-en-Jarez
  - Chu Strasbourg, Strasbourg
  - CHU de TOULOUSE, Toulouse
  - CHU de Tours - Hopital Trousseau, Tours
  - CHU NANCY - Hopital Brabois, Vandœuvre-lès-Nancy